CLINICAL TRIAL: NCT05477173
Title: Psychiatric Disorders Related to Children With Diabetes Mellitus
Brief Title: Psychiatric Disorders Related to Diabetes Mellitus Type 1 Among Children in Egypt
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Gellan Karamalllah Ramadan Ahmed, lecturer of neurology and psychiatry,faculty of medicine, Assiut University
Other Study IDs: diabetes children
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Diabetes Mellitus Type 1; Adolescents; Psychiatric Disorders
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: The Strengths and Difficulties Questionnaire (SDQ) Parent Version Parent : It consists of 25 questionnaires used to screen for behavioral problems in children aged 4-17 years. — screen by using psychometric scales
  Other Names: The Children's Alexithymia Measure (CAM) : The CAM comprises 14 components rated in a range of 0 to 3.Total scores can vary from 0 to 42, with higher numbers indicating more alexithymia; the Children's Sleep Habits Questionnaire (CSHQ-A) was used to assess sleeping difficulties.

SUMMARY:
Type 1 diabetes is the most common endocrine disorder in children and adolescents. It is characterised by a deficiency in insulin synthesis and requires daily insulin injections to manage glucose levels. Therefore, there are numerous medical approaches to its therapy, such as levels of glycosylated haemoglobin (HbA1c) as a marker of glycaemic control during the last 3 months and monitoring of blood glucose levels, influencing the mental health and the quality of life of the patient and family. Hens, the importance of the psychological adjustment to children and adolescents with type 1 diabetes besides insulin injection, adequate diet and regular exercise rises, in order to maintain stable psychological status and functional mental health, and prevent psychological disorders such as anxiety, depression and sleep disorders. Approaching the comorbidity in these children and adolescents starts with the diagnosis and with the health changes in all aspects.

ELIGIBILITY:
Inclusion Criteria:

1. Both boys and girls aged 6-12 years.
2. Willing of the parents or the caregivers to participate in the study.
3. Duration of type 1 DM of at least 1 year.

Exclusion Criteria:

1. Children with intelligence quotient below 70.
2. Children with history of substance use.
3. Children with another medical or neurological conditions.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with Diabetes Mellitus Type 1
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Measure frequency of sleep problems with diabetes mellitus type 1 | through study completion, an average of 1 year
Measures frequency of psychiatric problems with diabetes mellitus type 1 | through study completion, an average of 1 year

IPD SHARING:
Plan to Share IPD: Undecided